CLINICAL TRIAL: NCT06794593
Title: Effect Camostat for Kidney Protection in Chronic Kidney Disease
Acronym: CamKid
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EUCT 2023-508516-34-00; 2023-508516-34-00 (EU CTIS Number)
Record Dates: First submitted 2025-01-10; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Chronic Kidney Disease(CKD)
Keywords: CKD; Chronic Kidney Disease; Proteinuria; Camostat Mesylate; Serine Protease Inhibitor; Complement; ENaC; Epithelial Sodium Channel; Albuminuria; Proteaseuria
MeSH Terms: conditions — Renal Insufficiency, Chronic; Proteinuria; Albuminuria | interventions — camostat

STUDY DESIGN:
Intervention Model Description: This is a single-center, interventional, non-randomized, open-label pharmacodynamic study designed to evaluate the effects of Camostat Mesilate in patients with chronic kidney disease (CKD) and proteinuria compared to healthy controls. A total of 40 participants (20 CKD patients and 20 healthy controls matched by age and gender) will follow a standardized sodium diet (150 mmol/day) for 8 days. On the fifth day, participants will begin a 4-day course of oral Camostat (200 mg three times daily), while continuing the sodium-controlled diet. CKD patients will receive CM as an add-on to their standard treatment. Blood samples, 24-hour urine collections, home blood pressure measurements, and body composition monitoring will be performed at baseline, after 4 days on the diet, and after completing the Camostat treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chronic Kidney Disease patients (Experimental): Patients with chronic kidney disease. eGFR > 30 ml/min/1,73 m^2 and U-ACR > 300 mg/g.
  Interventions: Drug: Camostat Mesylate
- Healthy Controls (Experimental): Healthy males and females in good general health and with no significant medical conditions or chronic illness.
  Interventions: Drug: Camostat Mesylate

INTERVENTIONS:
Drug: Camostat Mesylate — Oral Camostat Mesylate 200 mg x 3 daily for 4 days.
  Other Names: Foipan

SUMMARY:
This clinical trial aims to evaluate the effects of Camostat Mesylate, a serine protease inhibitor, in patients with chronic kidney disease (CKD) and proteinuria. Proteinuria accelerates CKD progression and increases cardiovascular risks. By inhibiting serine protease activity and tubular complement activation, camostat may mitigate progressive kidney injury, potentially improving clinical outcomes.

This is an interventional, non-randomized, open-label pharmacodynamic trial that includes CKD patients with proteinuria and healthy controls. This approach has been chosen as the trial serves as a pilot study, aiming to investigate a novel treatment target in CKD patients. Including healthy controls allows a comparison of the effect of Camostat Mesilate on normal physiology versus CKD with proteinuria.

Participants will:

* Follow a standardized sodium diet of 150 mmol/day for 8 days.
* Receive oral Camostat Mesilate (200 mg thrice daily) for four days (day 5-8 on the diet).
* Provide blood and urine samples, record blood pressure, and undergo body composition measurements at baseline, during intervention, and at study completion.

The primary effect parameters are urine sodium and water excretion, body water content/weight, and home blood pressure. Secondary endpoints are tubular complement activation, urine protease activity, ENaC activation, 24-hour urine albumin excretion, and plasma concentrations of renin, angiotensin II, aldosterone, and NT-proBNP.

DETAILED DESCRIPTION:
Please refer to the protocol.

ELIGIBILITY:
Patients:

Inclusion criteria:

1. Age ≥ 18 years.
2. A clinical diagnosis of CKD of any course and meet the following criteria at screening:

   1. eGFR ≥ 30 ml/min/1.73m2
   2. U-ACR ≥ 300 mg/g.
3. Stable antihypertensive treatment 2 weeks before start of investigated medical drug (IMP) and maintain this treatment throughout the study.
4. Office blood pressure at the screening session should be >120/70 mmHg and <150/90 mmHg.
5. Capable of providing a signed informed consent and comply with study requirements.
6. Women with childbearing potential must have a negative pregnancy test (urine hCG) at spot urine at the screening visit and should use contraception during the study and until one week after completion of study treatment.

Exclusion criteria:

1. Treatment with Amiloride, Spironolactone, Aldosterone, or analogues.
2. Treatment with NSAIDs.
3. Hyperkalemia > 5.0 mmol/L at screening.
4. P-bilirubin > 25 umol/L at screening.
5. Ongoing cancer treatment.
6. Treatment with immunosuppressive therapy within 6 months prior to screening.
7. History of organ transplantation.
8. Evidence of current infection (CRP>50 or temperature > 38 C°).
9. Severe hepatic insufficiency classified as Child-Pugh C.
10. Breastfeeding.
11. Congestive heart failure NYHA class IV, unstable or acute congestive heart failure.
12. Recent cardiovascular events < 2 months prior to screening:

    1. Coronary artery revascularization.
    2. Acute stroke or TIA.
    3. Acute coronary syndrome.
13. Allergy or hypersensitivity to the IMP.
14. Addison's disease.
15. Gastric bypass operation.
16. Lactose intolerance since lactose serves as one of the inactive ingredients in the IMP.
17. Participation in other clinical trials within the last 30 days.

Healthy controls:

Inclusion criteria:

1. Age ≥ 18 years.
2. Good general health with no significant medical conditions or chronic illness (e.g., diabetes, hypertension, cardiovascular disease, autoimmune diseases, and cancer).
3. Normal kidney function and no proteinuria at screening:

   1. eGFR > 90 ml/min/1.73m2
   2. U-ACR < 30 mg/g
4. Office blood pressure at the screening < 140/90 mmHg.
5. Capable of providing a signed informed consent and comply with study requirements.

7. Women with childbearing potential* must have a negative pregnancy test (urine hCG) at spot urine at the screening visit and should use contraception during the study and until one week after completion of study treatment.

Exclusion criteria:

1. Treatment with any prescription medication except oral contraceptives.
2. Use of NSAIDs (Non-Steroidal Anti-Inflammatory Drugs)
3. Hyperkalemia > 5.0 mmol/L at screening.
4. P-bilirubin > 25 umol/L at screening.
5. Evidence of current infection (CRP>50 or temperature > 38 C°).
6. Breastfeeding.
7. History of substance abuse including alcohol.
8. Allergy or hypersensitivity to the IMP.
9. Gastric bypass operation.
10. Lactose intolerance since lactose serves as one of the inactive ingredients in the IMP.
11. Participation in other clinical trials within the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
24 h Urine sodium excretion (mmol/day) | At baseline (day 0), before treatment with IMP (day 5), and after completion of 4 days treatment with IMP (day 9).
Water excretion (L) | At baseline (day 0), before treatment with IMP (day 5), and after completion of 4 days treatment with IMP (day 9).
  24 h urine collection
Total Body Water (L) | At baseline (day 0), before treatment with IMP (day 5), and after completion of 4 days treatment with IMP (day 9).
  Measured by Body Composition Monistor
Home blood pressure | At baseline (day 0), before treatment with IMP (day 5), and after completion of 4 days treatment with IMP (day 9).

SECONDARY OUTCOMES:
Urine protease activity: zymography + protease activity | At baseline (day 0), before treatment with IMP (day 5), and after completion of 4 days treatment with IMP (day 9).
Tubular complement activation | At baseline (day 0), before treatment with IMP (day 5), and after completion of 4 days treatment with IMP (day 9).
  Urine C3a, MAC-sC5b-9, C3dg, MBL
Urine microvesicles: gammaENaC cleavage | At baseline (day 0), before treatment with IMP (day 5), and after completion of 4 days treatment with IMP (day 9).
Urine microvesicles: complement deposition | At baseline (day 0), before treatment with IMP (day 5), and after completion of 4 days treatment with IMP (day 9).
24 hours urine albumin excretion (mg/day) | At baseline (day 0), before treatment with IMP (day 5), and after completion of 4 days treatment with IMP (day 9).
Plasma concentration of renin, NT-proBNP, angiotensin II and aldosterone | At baseline (day 0), before treatment with IMP (day 5), and after completion of 4 days treatment with IMP (day 9).

CONTACTS AND LOCATIONS:
Overall Officials: Claus Bistrup, MD, Professor, Study Director — Department of Nephrology, Odense University Hospital, Denmark
Locations (1):
- Department of Nephrology, Odense University Hospital, Odense, Denmark

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-24): https://cdn.clinicaltrials.gov/large-docs/93/NCT06794593/Prot_SAP_000.pdf